CLINICAL TRIAL: NCT03190928
Title: Prospective Study of Clonal Evolution in Follicular Lymphoma
Brief Title: Clonal Evolution in Follicular Lymphoma
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170105; 17-C-0105
Record Dates: First submitted 2017-06-16; First posted 2017-06-19 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12-11

CONDITIONS: Follicular Lymphoma
Keywords: Disease Monitoring; Molecular Monitoring; Novel Biomarker Identification; Gene Expression Analyses; Watchful-Waiting; Natural History
MeSH Terms: conditions — Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with grades 1-2 or 3a follicular lymphoma (FL)

SUMMARY:
Background:

Follicular lymphoma is a type of cancer of the lymph nodes. Lab studies are important for cancer research. They help scientists better understand differences in the cancer biology of different patients. Researchers want to collect serial samples over time from people with follicular lymphoma to help them design future treatments.

Objective:

To collect a variety of samples from people with follicular lymphoma to study how these diseases progress and respond to treatment.

Eligibility:

Adults at least 18 years old who have been diagnosed with, but have not yet had any treatment for, follicular lymphoma.

Design:

Participants will be screened with medical history and physical exam. They will answer questions about daily functioning. They will have blood and urine tests. They may have scans and have tissue samples taken.

Participants will be monitored about every 4 months for up to 2 years. They will repeat screening tests. They will have a cheek swab. A small brush will be rubbed against the inside of the cheek to wipe off some cells.

Participants will have imaging scans about every 8 months for up to 2 years.

Participants may have a bone marrow aspiration and biopsy. The hipbone will be numbed with a small needle.

A needle will be put into the hipbone, and about 2 tablespoons of bone marrow will be taken out through the needle.

Participants will continue being monitored every 6 months for up to 5 years, then 1 time a year.

DETAILED DESCRIPTION:
Background:

* Follicular lymphoma (FL) is the second most common form of non-Hodgkin lymphoma and is incurable with standard first-line systemic therapy
* The clinical course of FL varies from slowly progressive over many years to a more rapid disease course that requires therapy shortly after diagnosis
* Early initiation of therapy does not improve survival, and asymptomatic patients are often managed with an initial period of watchful waiting
* Clinical prognostic indices predict survival, but cannot predict outcome for individual patients; biologic-based classifiers (gene-expression profiling and somatic mutational analyses) are more robust than clinical indices, but require prospective clinical validation from the time of diagnosis in the modern treatment era
* Paired samples linked to clinical information can lead to the discovery and/or validation of therapeutic targets for FL patients at the highest risk of early disease progression

Objective:

Characterize the molecular biology and clinical course of FL patients, and evaluate the time to treatment initiation for those patients who require first-line systemic therapy.

Eligibility:

* Follicular lymphoma (grade 1-2, 3a) with no evidence of histological transformation
* No previous cytotoxic, biologic or monoclonal antibody therapy for FL (previous radiation therapy permitted)
* Age greater than or equal to 18 years
* ECOG performance status of 0-2

Design:

* Patients with FL who meet all eligibility criteria will enroll on the study for expert monitoring of their disease, improved risk-stratification, and donation of tissue and cellular products for research. Patients will be monitored prospectively until they require second-line systemic treatment or the patient decides to withdraw from the study; untreated patients will be followed with clinic visits every 4 months for the first 2 years. After 2 years, protocol-specified visits will be increased to every 6 months until 5 years. After 5 years, protocol-specified visits will be annually until disease progression requiring first-line therapy.
* Patients without an indication for first-line systemic therapy at 2 years from initial study enrollment will be offered an optional biopsy of their lymph node and bone marrow.
* During first-line systemic therapy, patients can continue being monitored on this study for post-therapy clonal evolution. Protocol-specified visits after therapy will be every 6 months until 3 years. After 3 years, protocol-specified visits will be annually until disease progression requiring second-line therapy.
* Upon initiation of second-line therapy, if applicable, patients will move to survival follow-up only.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Histologically or cytologically confirmed follicular lymphoma (FL), grades 1-2, or 3a confirmed by the Laboratory of Pathology, NCI; patients who meet criteria for immediate initiation of systemic therapy are eligible
* Adequate tissue available from original diagnostic biopsy.

NOTE: If biopsy was >12 months prior to enrollment OR adequate tissue is not available, tissue biopsy may be optionally repeated unless such a biopsy is considered unacceptable risk to the patient. Patients without adequate tissue are eligible at the discretion of the PI.

- Must have disease that is measurable or evaluable on either computed tomography (CT) scans or FDG-positron emission tomography (FDG-PET) scans

NOTE: Since patients with FL may have lesions that wax and wane on imaging, the requirement for disease being measurable or evaluable can come from imaging taken at any time at or after diagnosis, the most recent imaging prior to enrollment does not need

to show measurable or evaluable disease.

- Age greater than or equal to 18 years

NOTE: Patients with the pediatric-type follicular lymphoma are usually <18 years of age, and often have a very different clinical course than patients with the adult-type of FL. Due to this difference in biology, children are excluded from this study.

- ECOG performance status <2 (Karnofsky >60%)

EXCLUSION CRITERIA:

* Previous history of diffuse large B-cell lymphoma or histologic transformation
* Any prior systemic treatment for lymphoma including cytotoxic chemotherapy, biologic therapy, and monoclonal antibody therapy (radiotherapy permitted); patients who have received chemotherapy, biologic therapy, hormonal therapy, or monoclonal antibody for other malignancies are potentially eligible provided that all of the following are true: a) that malignancy was not lymphoma, b) systemic therapy ended at least 3 years prior to the diagnosis of FL, and c) there is no evidence of active malignancy other than FL

NOTE: Initiation of first-line systemic therapy is allowed while on this trial; concurrent participation in first-line treatment clinical trials will be permitted.

* Patients who are HIV-positive
* Any second malignancy that requires active systemic therapy
* Any other (non-lymphoma) life-threatening disease
* Patients unable to provide informed consent (surrogates will not be used)
* Pregnant women are excluded from enrollment onto this study because the invasive procedures and/or sedation needed to perform them may cause unnecessary harm to the unborn fetus. In the event a woman becomes pregnant while on study, she will not be removed from the study; however, no follow-up invasive clinical or research procedures will be done that include unacceptable to risk to the patient and/or to the unborn fetus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 200 patients with pathologically-confirmed follicular lymphoma (grades 1-2, 3a) will be enrolled and screened for eligibility, and up to 80 eligible patients will receive active surveillance on this study for the purpose of expert monitoring of their disease, improved risk-stratification, and donation of tissue and cellular products for research.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-07-27 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Characteristics of treatment received (e.g., type, response, etc.) and molecular biology (e.g., pathology, histologic transformation) will be described | ongoing
  The types and frequency of each treatment will be reported.
Time to initiation of first-line systemic treatment (TTT1), defined as the number of days from study enrollment until the date of initiation of first-line systemic treatment | 2 years
  Number of days from study enrollment until the date of initiation of first-line systemic treatment will be reported.

SECONDARY OUTCOMES:
Progression-free survival | 2 years
  The number of days from initial diagnosis until date of first objective progression or death from any cause
Progression-free survival after first-line systemic treatment, defined as the number of days from diagnosis to objective disease progression after first-line systemic treatment | 5 years
  The number of days from diagnosis to objective disease progression after first-line systemic treatment or death from any cause
Progression-free survival from first active lymphoma treatment | 5 years
  The number of days from initiation of first-line systemic treatment to objective disease progression or death from any cause
Time to initiation of second-line systemic treatment | 5 years
  The number of days from study enrollment until the date of initiation of second-line systemic treatment
Overall survival (OS) | 10 years
  The number of days from initial diagnosis until death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Lakhotia, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request. @@@@@@All large scale genomic sequencing data will be shared with subscribers to dbGaP.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.@@@@@@Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.
Access Criteria: Genomic data are available once genomic data are uploaded per protocol GDS plan for as long as database is active.@@@@@@Genomic data are made available via dbGaP through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0105.html